CLINICAL TRIAL: NCT07141277
Title: GRANITE: Airsupra Effectiveness in the Real World A Retrospective Prevalent New-user Cohort Study to Describe Characteristics and Compare Effectiveness of Airsupra vs Albuterol, in Patients With Asthma Requiring Use of Rescue Therapy in a Real-world Setting in the United States
Brief Title: GRANITE: Airsupra Effectiveness in the Real World
Acronym: GRANITE
Status: Recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D6930R00007
Record Dates: First submitted 2025-07-11; First posted 2025-08-26 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Airsupra cohort: Eligible adults aged ≥18 years with asthma and at least one prescription for Airsupra
  Interventions: Other: None (Observational study)
- Albuterol cohort: Eligible adults aged ≥18 years with asthma and at least one prescription for albuterol
  Interventions: Other: None (Observational study)

INTERVENTIONS:
Other: None (Observational study) — Not applicable since it's an observational study.
  Other Names: Observational study

SUMMARY:
The GRANITE study aims to evaluate the effectiveness of Airsupra versus albuterol in reducing asthma exacerbation risk in a real-world US population.

ELIGIBILITY:
Inclusion Criteria:

* Patients with at least one prescription record (based on NDC or healthcare common procedure coding system [HCPCS] codes) of Airsupra (for Airsupra arm) or albuterol (for selected albuterol comparator arm) since January 2023
* Patients with an asthma indication (indicated by an ICD-10-CM code J45.xx) within the 12 months prior to the index date identified by at least one of the following Health Plan Employer Data Information Set (HEDIS) criteria:

At least one IP claim with asthma as the principal admission diagnosis, At least one ED/urgent care claim with asthma as the principal diagnosis, At least four outpatient claims with asthma as one of the listed diagnoses AND at least two claims for any asthma medications (including any rescue or maintenance medications) within the 12 months prior to the index date, At least four prescriptions for any asthma medications within the 12 months prior to the index date;

* Patients with at least one prescription record (based on NDC or HCPCS codes) of albuterol within the 12 months prior to the index date
* Patients aged ≥18 years on the index date
* Patients with ≥12 months of continuous insurance enrolment prior to and post index date

Exclusion Criteria:

* Patients with at least one medical claim with an ICD-10 code within the 12 months prior to the index date for the following chronic respiratory conditions or other systematic inflammatory diseases routinely treated with SCS: COPD, cystic fibrosis, pulmonary fibrosis, pulmonary arterial hypertension, bronchiectasis, respiratory tract cancer, hypereosinophilic syndrome, Churg-Strauss syndrome, eosinophilic pneumonia, Wegener's granulomatosis, allergic bronchopulmonary aspergillosis, obesity hypoventilation syndrome, hyperventilation syndrome, alpha-1 antitrypsin deficiency, primary ciliary dyskinesia, vasculitis collagen vascular disease, systemic lupus erythematosus, scleroderma, rheumatoid arthritis, Sjogren's syndrome, psoriatic arthritis, or inflammatory bowel disease (ulcerative colitis and Crohn's disease)
* Patients with maintenance OCS use within the 12 months prior to the index date, defined as use of OCS covering minimum 50% (6 months) in days' supply
* Airsupra patients with a concomitant SABA prescription record on the index date

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of a real-world adult population of asthma patients in a claims database using albuterol as rescue therapy.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2025-07-09 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Baseline demographics and clinical characteristics of patients receiving Airsupra and albuterol | Baseline period is 12 months prior to the index date
  Patient characteristics including demographics, clinical characteristics, asthma treatments, dosing, adherence to maintenance, asthma exacerbations, HCRU, and asthma severity defined per GINA will be described during the 12-month baseline period using descriptive statistics.
Severe asthma exacerbations | Follow-up period for each patient starts the day after the index date and ends at the earliest date of: end of data period,end of continuous enrolment(after 12 months),switch to albuterol(Airsupra cohort),Airsupra (albuterol cohort),or death.
  Number of patients with any severe asthma exacerbation and the rate of severe asthma exacerbation per person-year will be described during the follow-up period.

SECONDARY OUTCOMES:
Median time to first exacerbation | Follow-up period for each patient starts the day after the index date and ends at the earliest date of: end of data period,end of continuous enrolment(after 12 months),switch to albuterol(Airsupra cohort),Airsupra (albuterol cohort),or death.
  Time to first severe asthma exacerbation will be analyzed using the KM method and corresponding estimates of cumulative incidence over time will be plotted.
Total exposure for SCS and SCS bursts rates | Follow-up period for each patient starts the day after the index date and ends at the earliest date of: end of data period,end of continuous enrolment(after 12 months),switch to albuterol(Airsupra cohort),Airsupra (albuterol cohort),or death.
  Total exposure (days) for SCS, and SCS bursts rates will be described using summary statistics suitable for the distribution of the data.
Annualized exposure to Inhaled Corticosteroid (ICS) | Follow-up period for each patient starts the day after the index date and ends at the earliest date of: end of data period,end of continuous enrolment(after 12 months),switch to albuterol(Airsupra cohort),Airsupra (albuterol cohort),or death.
  Annualized exposure to ICS in μg/year fluticasone equivalents.
Annualized exposure to Systemic Corticosteroids (SCS) | Follow-up period for each patient starts the day after the index date and ends at the earliest date of: end of data period,end of continuous enrolment(after 12 months),switch to albuterol(Airsupra cohort),Airsupra (albuterol cohort),or death.
  Annualized exposure to SCS in mg/year prednisone equivalent.
Annualized exposure to ICS and SCS | Follow-up period for each patient starts the day after the index date and ends at the earliest date of: end of data period,end of continuous enrolment(after 12 months),switch to albuterol(Airsupra cohort),Airsupra (albuterol cohort),or death.
  Annualized total exposure to ICS and SCS the conversion factor of 5000 µg/day of inhaled budesonide to 10mg/day of oral prednisone will be used among Airsupra and the comparator albuterol cohort.

CONTACTS AND LOCATIONS:
Locations (1):
- AstraZeneca, Wilmington, Delaware, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org.
  Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/